CLINICAL TRIAL: NCT01709019
Title: A Phase I Randomized, Observer-Blinded, Dose-Ranging Study to Evaluate the Immunogenicity and Safety of an RSV-F Protein Nanoparticle Vaccine, With or Without Aluminum Adjuvant, and Co-administered With a Licensed Inactivated Influenza Vaccine, in Healthy Subjects ≥ 60 Years of Age.
Brief Title: RSV-F Vaccine and Influenza Vaccine Co-Administration Study in the Elderly
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novavax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NVX757.102
Record Dates: First submitted 2012-10-15; First posted 2012-10-17 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Respiratory Syncytial Virus (RSV)
MeSH Terms: interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group A (Experimental): Low dose RSV-F Vaccine with Adjuvant (Day 0); Seasonal TIV (Day 0 & Day 28)
  Interventions: Biological: Low dose RSV-F Vaccine with Adjuvant (Day 0); Seasonal TIV (Day 0 & Day 28)
- Group B (Experimental): Low dose RSV-F Vaccine without Adjuvant (Day 0); Seasonal TIV (Day 0 & Day 28)
  Interventions: Biological: Low dose RSV-F Vaccine without Adjuvant (Day 0); Seasonal TIV (Day 0 & day 28)
- Group C (Experimental): High dose RSV-F Vaccine with Adjuvant (Day 0); Seasonal TIV (Day 0 & Day 28)
  Interventions: Biological: High dose RSV-F Vaccine with Adjuvant (Day 0); Seasonal TIV (Day 0 & Day 28)
- Group D (Experimental): High dose RSV-F Vaccine without Adjuvant (Day 0); Seasonal TIV (Day 0 & Day 28)
  Interventions: Biological: High dose RSV-F Vaccine without Adjuvant (Day 0); Seasonal TIV (Day 0 & Day 28)
- Group E (Placebo Comparator): Placebo (Day 0 & Day 28); Seasonal TIV (Day 28)
  Interventions: Biological: Placebo (Day 0 & Day 28); Seasonal TIV (Day 0)

INTERVENTIONS:
Biological: Low dose RSV-F Vaccine with Adjuvant (Day 0); Seasonal TIV (Day 0 & Day 28) — 0.5mL IM injections
  Arms: Group A
Biological: Low dose RSV-F Vaccine without Adjuvant (Day 0); Seasonal TIV (Day 0 & day 28) — 0.5mL IM injections
  Arms: Group B
Biological: High dose RSV-F Vaccine with Adjuvant (Day 0); Seasonal TIV (Day 0 & Day 28) — 0.5mL IM injections
  Arms: Group C
Biological: High dose RSV-F Vaccine without Adjuvant (Day 0); Seasonal TIV (Day 0 & Day 28) — 0.5mL IM injections
  Arms: Group D
Biological: Placebo (Day 0 & Day 28); Seasonal TIV (Day 0) — 0.5mL IM Injections
  Arms: Group E

SUMMARY:
Up to 220 eligible subjects will be enrolled into one of five treatment groups. It is anticipated that some of the randomized study subjects may not complete the study; subjects who withdraw or are discontinued, will not be replaced. Randomization will be stratified by age (60 to <75 years and ≥ 75 years) in order to distribute the proportion of such persons in each age group equally across treatment groups.

Treatments will comprise a single IM dose of a placebo or RSV-F protein nanoparticle vaccine on Day 0, with concurrent IM immunization with a licensed inactivated influenza vaccine. A rescue dose of the licensed TIV will be provided to subjects in all groups except the placebo group on Day 28, the placebo group will receive saline. For each subject, study follow-up will span approximately one year from the first immunization (on Day 0) for all subjects.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females, ≥ 60 years of age, without symptomatic cardiopulmonary disease. Note that subjects who have any functional limitation or symptoms related to cardiac and/or pulmonary disease (including asthma or other episodic symptoms), or who receive ongoing therapy to control symptoms or functional limitation, are not eligible. The following are examples of subjects who may bear cardio-pulmonary diagnoses but who would remain eligible:

  1. Subjects on stable (no change in ≥ 2 months) therapy for findings (e.g., hypertension or hyperlipidemia) that are not associated with current symptoms or disability.
  2. Subjects who receive intermittent prophylaxis for risks associated with asymptomatic findings (e.g., antibiotic prophylaxis prior to dental procedures in a subject with asymptomatic mitral valve prolapse).
  3. Other clinically insignificant findings, not deemed to be associated with increased risk due to respiratory viral infections as determined by the Investigator.
* Free of other illnesses which are believed to increase the risk of influenza or influenza related complications including: diabetes mellitus, congenital or acquired blood dyscrasias, renal or hepatic dysfunction, and morbid obesity.
* Willing and able to give informed consent prior to study enrollment.
* Able to comply with study requirements.

Exclusion Criteria:

* Participation in research involving investigational product (drug / biologic / device) within 45 days before planned date of first vaccination and/or planned participation at any time during the study.
* History of a serious reaction to any prior vaccination or known allergy to constituents of licensed TIV (e.g., egg proteins).
* History of Guillain-Barré Syndrome within 6 weeks following a previous influenza vaccine.
* Receipt of any influenza vaccine within the preceding 3 months.
* Receipt of any vaccine in the 4 weeks preceding the study vaccination and planned receipt of a licensed vaccine any time prior to Day 56.
* Receipt of an RSV vaccine at any time.
* Any known or suspected immunosuppressive condition, acquired or congenital, as determined by medical history and/or physical examination.
* Chronic administration (defined as more than 14 continuous days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the administration of the study vaccine. An immunosuppressant dose of glucocorticoid will be defined as a systemic dose ≥10 mg of prednisone per day or equivalent. The use of topical, inhaled, and nasal glucocorticoids will be permitted provided these are not administered for diagnoses inconsistent with the inclusion criteria. The use of inhaled glucocorticoids, although typically not associated with system absorption, will generally indicate the presence of a diagnosis inconsistent with inclusion criteria 1 or 2.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the administration of the study vaccine or during the study.
* Acute disease at the time of enrollment (defined as the presence of a moderate or severe illness with or without fever, or an oral temperature >38.0°C on the planned day of vaccine administration).
* Known disturbance of coagulation.
* Suspicion or recent history (within one year of planned vaccination) of alcohol or other substance abuse.
* Any condition that in the opinion of the Investigator would pose a health risk to the subject if enrolled or could interfere with evaluation of the vaccine or interpretation of study results (including neurologic or psychiatric conditions deemed likely to impair the quality of safety reporting).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2012-10; Primary Completion 2013-07 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Assessment of Safety | Day 0 to Day 364
  Number (and percentage) of subjects with solicited local and systemic Adverse Events over the seven days post injection; all adverse events, solicited and unsolicited over 56 days post-first injection.
  Significant New Medical Conditions, Medically Attended Events and Serious Adverse Events will be collected for one year.
Immunogenicity as assessed by serum IgG antibody titers for the F-Protein antigen | Day 0 to Day 364
  Immunogenicity will be measured using derived / calculated endpoints based on:
  * Geometric mean titer (GMT)
  * Geometric mean ratio (GMR)
  * Seroconversion rate (SCR)
  * Seroresponse rate (SRR)

SECONDARY OUTCOMES:
Immunogenicity as assessed by serum HAI titers specific for the influenza antigens contained in the seasonal vaccine. | Day 0 to Day 56
  Immunogenicity will be measured using derived / calculated endpoints based on:
  * Geometric mean titer (GMT)
  * Geometric mean ratio (GMR)
  * Seroconversion rate (SCR)
  * Seroprotection rate (SPR)

CONTACTS AND LOCATIONS:
Overall Officials: D. Nigel Thomas, Ph.D., Study Director — Novavax, Inc.
Locations (4):
- United States (4):
  - Genova Clinical Research, Tucson, Arizona
  - Accelovance, Melbourne, Florida
  - Research Across America, Dallas, Texas
  - Jean Brown Research, Salt Lake City, Utah

REFERENCES:
- [Derived] Fries L, Shinde V, Stoddard JJ, Thomas DN, Kpamegan E, Lu H, Smith G, Hickman SP, Piedra P, Glenn GM. Immunogenicity and safety of a respiratory syncytial virus fusion protein (RSV F) nanoparticle vaccine in older adults. Immun Ageing. 2017 Apr 12;14:8. doi: 10.1186/s12979-017-0090-7. eCollection 2017. PMID 28413427
- See also: Novavax Homepage — http://www.novavax.com